CLINICAL TRIAL: NCT02901223
Title: Oncoplastic Breast Surgery Allow Tumor Resection With More Oncological Safety Than Standard Quadrantectomy With Nice Cosmetic Results and Better Quality of Life
Brief Title: The Impact of Oncoplastic Breast Surgery on the Oncological Safety and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Abdel-samii, Lecturer of general surgery, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB0006379
Record Dates: First submitted 2016-08-31; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Non Metastatic Breast Cancer
Keywords: Oncoplastic breast surgery; oncological safety; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quadrantectomy group (Active Comparator): 35 female patients with non metastatic breast cancer who had standard conservative breast surgery by general breast surgeons.
  Interventions: Procedure: Standard quadrantectomy
- oncoplastic group (Active Comparator): 35 female patients with non metastatic breast cancer who had oncoplastic techniques for tumor resection by well trained oncoplastic breast surgeons.
  Interventions: Procedure: oncoplastic breast surgery

INTERVENTIONS:
Procedure: Standard quadrantectomy — standard conservative surgery with no use of any plastic techniques
  Arms: Quadrantectomy group
Procedure: oncoplastic breast surgery — Integration of plastic techniques with oncological procedures
  Arms: oncoplastic group

SUMMARY:
The aim of this study is to asses the oncological safety of oncoplastic breast surgery, its impact on patient satisfaction and is it worthy for general breast surgeon to learn different oncoplastic techniques.

DETAILED DESCRIPTION:
This non randomized prospective trial was conducted on 70 female patients presented to our tertiary referral breast unit -Ain Shams University hospitals with non metastatic breast cancer during the period from September 2012 to September 2013. All of them signed an informed consent to share in this study that was approved in the ethical committee held on April 2012 - Ain Shams University. Our patients were divided into 2 equal groups: group A (35patients) who underwent standard quadrantectomy, group B (35 patients) who underwent oncoplastic surgery. In group A all quadrantectomies were done by general breast surgeons while in group B the oncoplastic procedures were done by well trained oncoplastic breast surgeons not assisted by plastic surgeons. The following data were reported in all cases including: age, family history, tumor size, volume and weight of the specimen, location of tumor, margin length, (primary tumor, regional nodes, metastasis) staging, molecular subtype and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1, 2 breast cancer
* Non metastatic breast caner
* Singing informed consent

Exclusion Criteria:

* Metastatic breast cancer
* Stage 3, 4 breast cancer
* Inflammatory breast cancer
* Multicentric/multifocal disease
* Ductal carcinoma in situ
* Patients older than 60 years
* History of breast surgery in oncoplastic group
* Co-morbidity in oncoplastic group
* Patients more than 60 years old

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Margins in all specimens measured in millimeters. | two years.
Patient satisfaction assessed using questionnaire. | Two years.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasser mohamed abdel-samii El Ghamrini, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided